CLINICAL TRIAL: NCT04086017
Title: Teaching Caregivers of Hospice Patients to Administer Reiki for Symptom Management and Caregiver Support: A Feasibility Pilot Study
Brief Title: Teaching Caregivers of Hospice Patients to Administer Reiki
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of COVID-19 we moved to a virtual format but older patients and caregivers were not open to a virtual format.
Sponsor: Ohio State University (Other)
Collaborators: OhioHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019B0544
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Hospice; Pain; Anxiety; Stress
Keywords: symptom management; Reiki therapy; self-care
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial: intervention and usual care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki teaching (Experimental): Reiki Master will perform the teaching and attunement process for Level 1 Reiki and teach the caregiver(s) how to complete a simple 10-minute Reiki session with the patient and a 10-minute self-Reiki session for the caregiver(s). The Reiki Master will explain that Reiki sessions can be given whenever the patient and caregiver feel it is appropriate, but sessions should be at minimum twice per 24-hour period for at least 10 minutes with at least two hours between sessions. Reiki sessions may be more frequent than twice per day and/or longer than 10 minutes. Self-Reiki sessions should be performed daily for at least 10 minutes but maybe more frequent and/or longer in length. Each family caregiver will receive a copy of the book. The patient and caregiver will wear a Holter monitor continuously for 48 hours beginning when the caregiver(s) are trained in Reiki to measure HRV, a valid measure for stress.
  Interventions: Other: Reiki therapy
- Usual care (No Intervention): Patients and caregivers will complete all measures expected of the intervention cohort including daily symptom checklist for 10 days. The patient and caregiver will wear a Holter monitor for the first 48 hours of study participation to measure heart rate variability (HRV), a valid measure for stress. The patient and/or caregiver may opt out of the Holter monitor if requested and still participate in the rest of the study.

INTERVENTIONS:
Other: Reiki therapy — Reiki is a complementary health approach where trained providers place their hands lightly on or just above a person, in discrete positions, with the goal of facilitating the person's own healing response. A Reiki practitioner will perform the initial teaching and instruct the caregivers how to perform a simple 10-minute Reiki and self-Reiki session.
  Arms: Reiki teaching

SUMMARY:
Being a family caregiver for a patient at the end of life is both rewarding and stressful. When the end of life is nearing, caregivers may be unsure of how to help their family member. Reiki, a light touch energy therapy has been shown to increase relaxation and improve sleep quality, and decrease pain, anxiety, depressive symptoms, and medication use in both hospitalized and community-dwelling adults. This feasibility study is designed to evaluate whether teaching caregivers is feasible in addition to evaluating any benefit to FCGs and patients.

DETAILED DESCRIPTION:
The time a patient and family caregiver (FCG) spend together in a patient's final days is filled with emotion. Patients may turn inward and be filled with peace, or they may be bothered by symptoms. Caregivers often experience feelings of helplessness and anticipatory grief. Learning and providing a skill such as Reiki may give caregivers a way to help the patient with symptoms while at the same time feeling useful. Patient and caregiver closeness may be enhanced. Reiki has been shown to be helpful with symptoms such as pain, anxiety, depression, fatigue, and others. However, teaching caregivers of terminal hospice patients, Reiki has not been studied. The knowledge gained from this feasibility study will guide future interventions aimed at the comfort of hospice patients and FCGs.

Approximately 1.49 million Medicare beneficiaries received hospice care during 2017, and most had a FCG. During the final days or weeks, FCGs are unsure of what do or how to best help the patient when everyday caregiving actives such as physical care or nutrition are not required or no longer desired by the patient. Caregiver symptoms of depression, anxiety, or anticipatory grief increase toward the end of life along with increased patient symptoms. Having a specific skill to help the patient with symptoms or simply to show care and provide touch may empower FCGs and improve the quality of life for both caregivers and patients.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for the study if they are

* ≥ 18 years old
* receiving hospice at home.

Caregivers will be eligible if they are

* ≥ 18 years old,
* willing to complete measures, and if they are randomized to the Reiki group
* willing to learn Reiki therapy, provide at least two Reiki therapy sessions with the patient of at least 10 minutes twice per day with at least two hours between sessions and complete one 10-minute self-Reiki session per day. Two caregivers may participate in the study.

Exclusion Criteria:

Patients will be excluded if:

* they have a diagnosis of atrial fibrillation
* they have an active pacemaker, or
* death is expected in less than two weeks.

Caregivers will be excluded if they

* cannot understand or speak English
* have severe, uncorrected hearing loss
* have self-reported uncontrolled atrial fibrillation
* have a self-reported diagnosis of dementia
* have a self-reported psychiatric disorder (bipolar disorder, schizophrenia)
* are unwilling or unable to complete measures (both groups) or perform Reiki and self-Reiki (intervention cohort).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Establish successful enrollment of patient-caregiver dyads | 10 days
  Successful enrollment will be measured by the number of dyads enrolled versus those approached
Establish successful completion of patent-caregiver dyad data collection | 10 days
  Successful completion of data collection will be measured by the number of dyads who complete all data collection surveys from dyads enrolled

SECONDARY OUTCOMES:
Change in heart rate variability measured using a heart rate monitor | Day 1 and 2
  Explore heart rate variability as a measure of stress using a heart rate monitor in end-of-life patients and their caregivers
Explore family caregiver feelings related to Reiki through the System usability Scale (modified) | Day 11
  Explore family caregiver feelings related to Reiki by having caregivers complete the System Usability Scale (modified) at the end of the 10 day intervention period. The System Usability Scale is a 13 item survey that measures whether respondents thought that learning Reiki went well, was understandable, and if they were confident using Reiki. Each item is answered by circling an answer on a Likert scale from "strongly disagree" to "strongly agree."
Explore family caregiver feelings related to Reiki through the Reiki Experience Questionnaire (Reiki-EQ) | Day 11
  Explore family caregiver feelings related to Reiki by having caregivers complete the Reiki-EQ at the end of the 10 day intervention period. This questionnaire is a combination of Likert responses as well as optional an area for participants to write additional information if they would like. This questionnaire assesses what the participants thought about learning and providing Reiki.
Compare daily symptoms between patients in the intervention and usual care group | Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10
  Examine and describe changes in 6 symptoms daily using the Daily Symptom Severity Assessment (SSA). The SSA measures 6 symptoms (pain, anxiety, shortness of breath, nausea, sleep, and sense of inner peace/happiness) using a visual analog scale
Compare symptoms between patients in the intervention and usual care group | Days 0 and 11
  Examine and describe symptom profiles, present illness, and co-morbidities of patients using the Rotterdam Symptom Checklist. The Rotterdam Symptom Checklist is a list of 30 common symptoms. Following each symptom is a Likert scale with four choices ranging from "not at all" to "very much."
Compare daily symptoms between caregivers in the intervention and usual care group | Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10
  Examine and describe changes in 6 symptoms daily using the Daily Symptom Severity Assessment (SSA). The SSA measures 6 symptoms (pain, anxiety, shortness of breath, nausea, sleep, and sense of inner peace/happiness) using a visual analog scale
Compare symptoms between caregivers in the intervention and usual care group using the Rotterdam Symptom Checklist | Days 0 and 11
  Examine and describe symptom profiles, present illness, and co-morbidities of caregivers using the Rotterdam Symptom Checklist. The Rotterdam Symptom Checklist is a list of 30 common symptoms. Following each symptom is a Likert scale with four choices ranging from "not at all" to "very much."
Compare symptoms between caregivers in the intervention and usual care group using the PROMIS-43 Symptom Profile | Days 0 and 11
  Examine and describe symptom profiles of family caregivers using the Patient Reported Outcomes Measurement Information System (PROMIS-43). The PROMIS-43 asks 6 questions within each of 7 symptom domains (physical function, anxiety, depression, fatigue, sleep disturbance, social activities, and pain interference) as well as a pain intensity score from 0 to 10. Questions in symptom domains are scored on a 5 level Likert score from "not at all" or "never" to "very much" or "always." Scores on this measure are totaled with a lower score indicating a better ability to function.
Change in daily patient symptoms as measured by the daily Symptom Severity Assessment. | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10
  Explore the patient symptoms within the intervention and usual care groups as measured by the daily Symptom Severity Assessment (SSA) over the study period. The SSA measures 6 symptoms (pain, anxiety, shortness of breath, nausea, sleep, and sense of inner peace/happiness) using a visual analog scale. Changes will be assessed within the intervention and usual care groups.
Change in patient symptom profile as measured by the Rotterdam Symptom Checklist. | Days 0 and 11
  Explore the patient symptoms within the intervention and usual care groups as measured by the Rotterdam Symptom Checklist. Examine and describe symptom profiles, present illness, and co-morbidities of patients using the Rotterdam Symptom Checklist. The Rotterdam Symptom Checklist is a list of 30 common symptoms. Following each symptom is a Likert scale with four choices ranging from "not at all" to "very much."
Change in caregiver daily symptoms as measured by the daily Symptom Severity Assessment. | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10
  Explore the caregiver symptoms within the intervention and usual care groups as measured by the daily Symptom Severity Assessment (SSA) over the study period. The SSA measures 6 symptoms (pain, anxiety, shortness of breath, nausea, sleep, and sense of inner peace/happiness) using a visual analog scale. Changes will be assessed within the intervention and usual care groups.
Change in caregiver symptom profile as measured by the Rotterdam Symptom Checklist. | Days 0 and 11
  Explore the caregiver symptoms within the intervention and usual care groups as measured by the Rotterdam Symptom Checklist. Examine and describe symptom profiles, present illness, and co-morbidities of patients using the Rotterdam Symptom Checklist. The Rotterdam Symptom Checklist is a list of 30 common symptoms. Following each symptom is a Likert scale with four choices ranging from "not at all" to "very much."
Change in caregiver symptom profile as measured by PROMIS-43. | Days 0 and 11
  Explore the caregiver symptoms within the intervention and usual care groups as measured by Patient Reported Outcome Measurement Information System (PROMIS) symptom questionnaire over the study period. The PROMIS-43 asks 6 questions within each of 7 symptom domains (physical function, anxiety, depression, fatigue, sleep disturbance, social activities, and pain interference) as well as a pain intensity score from 0 to 10. Questions in symptom domains are scored on a 5 level Likert score from "not at all" or "never" to "very much" or "always." Scores on this measure are totaled with a lower score indicating a better ability to function.

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Thrane, PhD, RN, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University College of Nursing, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No